CLINICAL TRIAL: NCT05629494
Title: Effect of Non-steroidal Anti-inflammatory Drugs on Serum Prostate Specific Antigen Level
Brief Title: Anti-inflammatory Drugs and Serum Prostate-Specific Antigen Test
Acronym: ADAPT-PSA
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Albany Medical College (Other)
Responsible Party: Principal Investigator, Badar M. Mian, Professor of Urology, Albany Medical College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6587
Record Dates: First submitted 2022-09-03; First posted 2022-11-29 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Prostate Cancer; Prostate Inflammation; PSA
Keywords: Prostate-specific antigen; PSA test; Prostate biopsy; non-steroidal anti-inflammatory drugs NSAIDS
MeSH Terms: conditions — Prostatic Neoplasms; Prostatitis | interventions — Ibuprofen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Repeat serum PSA test (Active Comparator): Repeat PSA test at 6 (± 1) weeks, without any treatment
  Interventions: Diagnostic Test: PSA test
- Treatment with NSAIDS (Experimental): Treatment with Ibuprofen 400 mg, 3 times per day, then repeat PSA test at 6 (± 1) weeks
  Interventions: Drug: Ibuprofen 400 mg, TID; Diagnostic Test: PSA test

INTERVENTIONS:
Drug: Ibuprofen 400 mg, TID — Participants will receive Ibuprofen 400 mg 3 times per day for 10 days.
  Other Names: Motrin
  Arms: Treatment with NSAIDS
Diagnostic Test: PSA test — PSA test will be repeated in 6 weeks

SUMMARY:
Prostate cancer is the most frequently diagnosed cancer in men in the Unites States. Nearly 1 million prostate biopsy procedures are performed in the United States annually and elevated prostate-specific antigen (PSA) level is the primary reason for prostate biopsy in > 90% of cases. However, at the PSA levels which trigger prostate biopsy, often no cancer is found in prostate biopsy specimens. PSA test can be elevated due to reasons other than cancer such as inflammation or natural variation in the level. Investigators plan to treat men with elevated PSA level with over the counter anti-inflammatory medications (ibuprofen, naproxen) to see if the PSA level will decrease to an acceptable level.

DETAILED DESCRIPTION:
It's known that PSA level can be elevated due to reasons other than prostate cancer including benign prostatic hypertrophy, prostatitis or other urinary tract infections, non-infectious inflammation, and physiologic variation over time. Consequently, nearly 50% of prostate biopsy procedures performed due to elevated PSA level do not yield any cancer , but still expose the patients to the risks of the procedure related complications (discomfort/pain, anxiety, bleeding, infection, and cost). Thus, measures to improve the reliability of PSA test, and potentially avoiding unnecessary procedures, are of significant importance to the patient and healthcare system.

It is common practice to check PSA level annually. PSA test results can vary over time, either due to the imprecision in the analysis and/or due to the biologic variability. This can result in an apparent rise in PSA level when no clinically meaningful rise had occurred. Its estimated that the average lab variation in PSA was approximately 6% and the average biologic variation about 14%. This, it is recommended that isolated elevation in PSA level should be confirmed after several weeks, and before proceeding with further interventions, including prostate biopsy.

Sub-clinical, histologic Inflammation (presence of inflammatory cells) within the prostate tissue and its effect on PSA level has been reported in various settings. In two population-based studies, men who were regularly using over the counter (OTC) nonsteroidal anti-inflammatory drugs (NSAIDs, e.g ibuprofen, naproxen) had lower PSA levels compared to non-users.

Currently, two strategies are utilized in clinical practice to ensure that the PSA level is truly elevated:

1. Repeat PSA test after several weeks or
2. A short course of OTC NSAIDs, and then repeat PSA test

Investigators propose to conduct a randomized study to determine the effect of NSAIDs on PSA level compared to the biologic variations in PSA level noted upon repeat testing.

ELIGIBILITY:
Inclusion Criteria:

* Male patients age between 18-80 years old with a screening PSA > 3 ng/ml being considered for additional diagnostic testing (e.g., MRI, biopsy)
* Normal digital rectal examination within the past two years. A documented normal digital rectal examination by another physician or advanced practice provider (NP, PA, etc) is acceptable.
* No clinical symptoms concerning for acute urinary tract infection (e.g. dysuria, malodorous urine, positive urine culture)

Exclusion Criteria:

* History of hypersensitivity or allergy to ibuprofen or NSAIDs.
* History of peptic ulcer disease, GI bleeding or NSAIDs induced GI adverse events
* Known bleeding disorders
* Known severe chronic kidney disease: eGFR < 30 mL/min/1.73 m2
* Heart failure, significant heart disease
* Poorly controlled hypertension
* Active urinary tract infections or bacteriuria
* Concomitant use of 5-alpha reductase inhibitors (finasteride, dutasteride) unless patient has been taking it for at least 6 months
* Known prostate cancer or underwent prostate MRI or biopsy in the last year
* Urinary tract instrumentation in the past 6 weeks (catheter, cystoscopy)
* Concomitant anti-inflammatory or steroidal drugs
* Concomitant dual-antiplatelet or anticoagulant therapy use except aspirin 81 mg alone
* Know history of severe liver disease determined by abnormal liver function tests (elevated AST or ALT > 3X ULN based on exiting history or labs)
* Any other medical contraindication to NSAIDs

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Estimated)
Dates: Start 2022-09-27 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Difference in the extent of changes in PSA level between the study groups | 6 weeks
  Difference in PSA levels, within and between groups
Participants with change in PSA level to below the age-specific PSA threshold | 6 weeks
  To determine if changes in PSA level were sufficient to avoid intervention

SECONDARY OUTCOMES:
Determine the incidence of acute kidney injury following a short course of ibuprofen | 1 year
  To determine if the treatment and PSA changes correlates with change in urinary symptoms
Durability of the change in PSA levels | 1 to 1.5 year
  Serial PSA levels will be examined to determine whether the change in PSA level is transient or durable
Changes in voiding symptoms as measured by the International Prostate Symptom Score | 3-12 months
  Patient reported symptom score, ranging from 0-35 (higher score=worse outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Badar Mian, MD, Principal Investigator — Albany Medical College; Jay Raman, MD, Principal Investigator — Penn State Health; Scott Eggener, MD, Principal Investigator — University of Chicago
Locations (3):
- United States (3):
  - University of Chicago Medical Center, Chicago, Illinois
  - Albany Medical Center, Albany, New York
  - Penn State-Hershey Medical Center, Hershey, Pennsylvania

IPD SHARING:
Plan to Share IPD: No